CLINICAL TRIAL: NCT05835154
Title: Improving Advance Care Planning Around Mobility Needs Among Patients With Sarcoma
Brief Title: A Checklist (Advanced Care Planning) for The Assessment of Mobility Needs in Patients With Sarcoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RG1123026; NCI-2022-09848 (Other: CTRP (Clinical Trial Reporting Program)); 11174 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2023-04-17; First posted 2023-04-28 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Sarcoma; Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Restraint, Physical; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (advanced care planning checklist) (Experimental): FIELD TEST: Participants complete the Advance Care Planning (ACP) Mobility Checklist on study. Participants complete questionnaires at baseline and after completing the checklist intervention and undergo interview on study. Participants medical records are also reviewed.
  Interventions: Behavioral: Assessment; Other: Questionnaire Administration; Other: Interview; Other: Electronic Health Record Review

INTERVENTIONS:
Behavioral: Assessment — Complete checklist
  Other Names: Assess
Other: Questionnaire Administration — Complete questionnaires
Other: Interview — Undergo semi-structured feedback interview
Other: Electronic Health Record Review — Review of medical records

SUMMARY:
This trial tests how well the advanced care planning around mobility needs checklist tool works to assess future mobility needs in patients with sarcoma. Gathering information about sarcoma patients that have had surgery to either save or remove a limb may help doctors learn more about a patient's mobility needs. Using an advance care planning mobility needs assessment may help improve the quality of life in patients with sarcoma by helping them plan for their future mobility needs.

DETAILED DESCRIPTION:
OUTLINE:

FIELD TEST: Participants complete the advance care planning (ACP) Mobility Checklist on study. Participants complete questionnaires at baseline and after completing the checklist intervention and undergo interview on study. Participants' medical records are also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS: Age 18 years of age or older.
* PATIENTS: English speaking
* PATIENTS: Able to provide informed consent
* PATIENTS: Have access to a computer or other device to fill out the online checklist
* PATIENTS: Have had either limb salvage or amputation surgery for sarcoma within the last 6 months OR have metastatic (stage IV) sarcoma and are in active treatment.
* CAREGIVERS: Age 18 years of age or older
* CAREGIVERS: English speaking
* CAREGIVERS: Able to provide informed consent
* CAREGIVERS: Have access to a computer or other device to fill out the online checklist
* CAREGIVERS: The person (family member or friend) whom the patient indicates being an informal caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility, as measured by the number of subjects accrued to the study | At enrollment
  The number of participants accrued during the recruitment period.
Feasibility, as measured by the number of subjects to complete the intervention | Through study completion, up to 4 weeks
  The number of participants to complete the intervention.
Acceptability of the intervention: Acceptability E-Scale | After completion of intervention (+ 1 week)
  The Acceptability E-Scale is a 6-item scale, scored on a 5-point Likert scale (e.g., 1=very difficult; 5= very easy), with previously demonstrated good internal consistency (Cronbach's alpha=.76), with higher values indicating higher levels of acceptability.
Usability: System Usability Scale (SUS) | After completion of intervention (+ 1 week)
  Usability of the ACP Mobility Checklist will be assessed among patients using the System Usability Scale (SUS). The SUS is a 10-item scale, scored on a 5-point Likert scale (1=strongly disagree; 5=strongly agree), with higher values indicating higher levels of usability.
Acceptability: Satisfaction with the intervention | After completion of intervention (+ 1 week)
  Satisfaction with the intervention will be assessed with a single, 10-point Likert scale item assessing how satisfied participants are with the intervention (1= not at all satisfied, 10 = extremely satisfied). Higher values indicate higher ratings of satisfaction.

SECONDARY OUTCOMES:
Change in planning for mobility needs | From baseline to after completion of intervention (+ 1 week)
  Will be measured by asking participants seven items about what mobility needs they have planned for (e.g., assistance with home environment, toileting, dressing, etc.) (yes/no). Total scores can range from 0 to 7, with higher values indicating higher rates of understanding and awareness.
Change in functional status | From baseline to after completion of intervention (+ 1 week)
  Functional status will be measured using the PROMIS Cancer Function Brief, which is a validated 12-item scale scored on a 5-point Likert scale, with higher scores indicating better functioning.
Change in patients' engagement in clinical conversations (present/absent) with specialist providers | From baseline to after completion of intervention (+ 1 week)
  Engagement in clinical conversations (present/absent) with providers will be measured with four questions asking patients if they have had an interaction or consult with a physical therapist, occupational therapist, speech language pathologist, and/or rehabilitation physician (yes/no). Total scores can range from 0 to 4, with higher values indicating higher rates of engagement in clinical conversations with specialist providers.
Change in discussion of advance directives | From baseline to after completion of intervention (+ 1 week)
  This will be measured using our previously utilized 8-item measure of discussing end-of-life care, living will, healthcare proxy, and do-not-resuscitate orders with family and doctor (all yes/no questions).
Change in completion of advance directives | From baseline to after completion of intervention (+ 1 week)
  This will be assessed by asking patients whether they have completed a Do Not Resuscitate order (DNR), living will, or identified a Health Care Proxy (HCP). All yes/no questions.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Shen, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No